CLINICAL TRIAL: NCT05436808
Title: Prospective Pilot Study of Partial Chest Wall Radiation Therapy (PCWRT) for Positive or Close Margins After Modified Radical Mastectomy for Lymph Node-Negative Breast Cancer
Brief Title: Partial Chest Wall Radiation Therapy After Surgery for Lymph Node Negative Breast Cancer
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No eligible participants identified
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Alexander Stessin, Associate Professor of Medicine, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBU-PCWRT-BREAST
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer; Breast Cancer Female; DCIS; Stage II Breast Cancer; Stage I Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Radiation Treatment (Experimental)
  Interventions: Radiation: Partial Chest Wall Radiation Therapy

INTERVENTIONS:
Radiation: Partial Chest Wall Radiation Therapy — Patients will receive radiation therapy (30 Gray in 5 fractions) to the affected chest wall, delivered on consecutive days or every other day

SUMMARY:
The standard treatment for breast cancer when cancer cells were found near or within the margins of the tissue that is removed during breast surgery, is radiation of the entire chest wall. This may be considered overtreatment since the only reason for doing so is that cancer cells were near or in the margins of the breast tissue that was removed. In this study, the amount of radiation treatment will be limited to the area where the remaining cancer cells were found after surgery.

The purpose of this study is to find out if partial chest wall radiation therapy is as good as whole chest wall radiation therapy in reducing the risk of breast cancer cancer coming back.

ELIGIBILITY:
Inclusion Criteria:

* DCIS or stage T1 or T2 invasive breast cancer, lymph node negative
* Must have undergone mastectomy
* Presence of cancer cells on or close to surgical margins
* Negative pregnancy test for women
* Must receive radiation at Stony Brook University Hospital

Exclusion Criteria

- Received prior radiation to are to be irradiated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Breast cancer recurrence | 5 years
  Number of patients with recurrent breast cancer
Acute toxicity | 3 months
  Frequency of radiation-related adverse events
Delayed toxicity | 5 years
  Frequency of radiation-related adverse events
Surgical complications | 5 years
  Number of patients with surgical complications

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Stessin, MD PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook Cancer Center, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No